CLINICAL TRIAL: NCT03606746
Title: A Phase 2 Prospective, Multi-center, Open-label Trial to Assess the Safety & Efficacy of Cellular Immunotherapy With MDR-103 for Induction of Mixed Chimerism & Immune Tolerance in Past Recipients of HLA Zero-mismatch, LD Kidney Transplants
Brief Title: Cellular Immunotherapy for Immune Tolerance in Past Recipients of HLA Zero-mismatch, Living Donor Kidney Transplants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Medeor Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDR-103-L2K
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplant Rejection
Keywords: Kidney Transplant; Kidney Failure; Anti-rejection therapy; Living Donor; HLA-matched; Hematopoietic Stem Cells (HSC); CD34+; CD3+; T cells; Cellular Therapy; Immunotherapy; Immunosuppression
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Arm (Experimental): A low-dose Total Lymphoid Irradiation (TLI) and anti-thymocyte globulin (ATG) combined with a single IV infusion of MDR-103 and standard anti-rejection medications in past recipients of HLA Zero-mismatch living donor kidney transplants.
  Interventions: Biological: MDR-103

INTERVENTIONS:
Biological: MDR-103 — MDR-103 Enriched CD34+ hematopoietic stem cells and defined dose of CD3+ T-cells

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of cellular immunotherapy with MDR-103 for induction of functional immune tolerance in past recipients of human leukocyte antigen (HLA)-matched, living donor kidney transplants.

DETAILED DESCRIPTION:
Currently, patients receiving a transplanted kidney are required to take life-long immunosuppressive medications to prevent rejection of the transplanted kidney. These medications carry substantial side effects. In addition, these medicines often do not completely control damage to the kidney from the recipients' immune system, ultimately causing the kidney to fail.

Medeor Therapeutics is developing a novel cell-based therapy to reprogram the past recipients' immune system to accept the transplanted kidney without the concurrent need for long term use of immunosuppressive drugs.

The purpose of the current Phase 2 study is to demonstrate the efficacy and safety of MDR-103 for the induction of transplant immune tolerance in a prospective, multicenter clinical trial. MDR-103 is intended to induce mixed lymphohematopoietic chimerism and donor specific immune tolerance in order to preserve transplant kidney function, avert transplant kidney rejection, and eliminate the cumulative and serious side effects associated with immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

Recipient Inclusion Criteria:

* Past recipient of a first kidney allograft from an HLA-matched, living related donor
* Age ≥18 and ≤70 years
* Single solid organ recipient (kidney only)
* ABO compatibility with donor

Donor Inclusion Criteria:

* HLA-matched first degree (parent, child or sibling) or second-degree (child of a sibling, half sibling) relative of the prospective recipient participant
* Age ≥18 and ≤70 years
* Past living related kidney donor, and capable of undergoing G-CSF mobilization and apheresis of hematopoietic cells

Exclusion Criteria:

Recipient Exclusion Criteria:

* Underlying kidney disease with a high risk of disease recurrence in the transplanted kidney
* Baseline positive donor-specific anti-HLA antibody testing
* Is taking immunosuppressive therapy
* Evidence of prior hepatitis B (HBV) or hepatitis C (HCV)

Donor Exclusion Criteria:

* History of autoimmune disorders
* History of type 1 or type 2 diabetes mellitus
* Tests confirmed positive for human immunodeficiency virus (HIV), HBV, HCV
* History of infection with Zika virus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Persistent Mixed Chimerism | At 6 months post initiation of anti-thymocyte globulin (ATG) conditioning therapy
  The primary efficacy endpoint is the proportion of subjects achieving persistent mixed chimerism in MDR-103 treated recipients of past HLA zero-mismatch living donor kidney transplants.
  Persistent Mixed Chimerism - is defined as at least 6 months of persistent WBC mixed chimerism consisting of at least 5% donor cells in whole blood or in at least one WBC lineage (CD3+ T cells, CD33+ myeloid cells, CD19+ B cells, and/or CD56+ NK cells).

IPD SHARING:
Plan to Share IPD: Undecided